CLINICAL TRIAL: NCT03085264
Title: Implementing 30-day Post- Discharge Community Health Worker Pairings for Patients at High-Risk for Readmission (C-CAT Study)
Brief Title: Community Health Worker Care Transitions Study
Acronym: CCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Carter, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017A050810
Record Dates: First submitted 2017-03-14; First posted 2017-03-21 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Hospitalism
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker (Experimental): Patients are paired with community health workers for 30 days after hospital discharge to assist with patient care
  Interventions: Behavioral: Community Health Worker
- Usual Care (No Intervention): Patients are not paired with community health workers for 30 days after hospital discharge to assist with patient care

INTERVENTIONS:
Behavioral: Community Health Worker — Community Health Workers calls, texts and visits patient to support them in pre-established care plans as well as medication compliance/appointment attendance
  Arms: Community Health Worker

SUMMARY:
This study focuses on pairing community health workers (CHWs) with patients that are high risk for readmission prior to hospital discharge in order to assess differences in hospital readmission rates, ED visits, patient satisfaction and provider satisfaction as compared to patients without community health worker pairings at discharge.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of 1200 adult patients admitted to internal medicine units that will examine the effectiveness of pairing patients that are high risk for readmission with community health workers at the time of hospital discharge on hospital readmission rates, emergency room visits, adherence to post-discharge medical appontments, and satisfaction with care. During this study, community health workers will partner with patients for 30 days after discharge from the hospital to address barriers to care via phone contacts, home visits, and accompanying patients to medical appointments/other non-clinical supportive care.

AIM 1) Determine if patients randomly assigned to the intervention group have lower rates of hospital readmission than the control group at the end of the intervention.

Hypothesis 1.1 Study participants in the intervention group will have lower rates of post-discharge thirty day readmission than the study participants in the control group at the end of the intervention.

AIM 2) Determine if patients randomly assigned to the intervention group will have less emergency room visits than the control group at the end of the intervention

Hypothesis 2.1 Study participants in the intervention group will have less emergency room visits than the study participants in the control group at the end of the intervention.

AIM 3) Determine if patients randomly assigned to the intervention group have more adherence to post-discharge appointments that study group participants in the control group at the end of the intervention

Hypothesis: 3.1 Study participants in the intervention group will have higher rates of attendance at post-discharge medical appointments than the study participants in the control group at the end of the intervention.

AIM 4) Determine if patients randomly assigned to the intervention group have higher levels of patient psychosocial support and satisfaction with post-discharge care than the control group

Hypothesis 4.1: Study participants in the intervention group will have higher levels of patient psychosocial support and satisfaction with post-discharge care than the study participants in the control group at the end of the intervention.

AIM 5) Determine if Primary Care Physicians of patients randomly assigned to the intervention group have higher levels of satisfaction with post-discharge care than Primary Care Providers of patients in the control group

Hypothesis 5.1: Primary Care Physicians of patients randomly assigned to the intervention group have higher levels of satisfaction with post-discharge care than Primary Care Providers of patients in the control group

After reviewing the fact sheet and consenting to enrollment by signing the informed consent form, patients will randomized to the intervention or control groups of the study.

STUDY PROCEDURES

Intervention Arm Group:

Patients randomized to the intervention group will be paired with community health workers prior to discharge from the hospital and patient- centered program goals will be established. A patient questionnaire (10-15 minutes) will be administered to intervention study participants by a study coordinator prior to discharge. A chart review will be performed for all intervention group participants by study coordinators prior to patient discharge. Patient-CHW pairings will continue for thirty days post-discharge and will include phone contacts, home visits, accompanying patients to medical appointments and other non-clinical supportive care. Both intervention group participants and primary care providers (PCPs) of intervention study participants will complete questionnaires 30-60 days after hospital discharge to assess certain patient ( 10 minute questionnaire; via phone) and primary care provider ( 5 minute questionnaire via email) perceptions (Please see Aim 4 and Aim 5). CHWs will document patient encounters in a REDCap database and complete patient care notes in EPIC. All intervention study participants readmitted within thirty days of prior discharge will be administered a readmission questionnaire by study coordinators. A chart review for readmitted study participants will also be performed by study staff. A REDCap database will be used to store all questionnaire and chart review data. Readmission rates, ED visits, PCP appointment compliance, patient/ PCP will be tracked.

Control Arm Group:

Those randomized to the control group will receive usual care without a community heath worker pairing. A patient questionnaire (10-15 minutes) will be administered to intervention study participants by a study coordinator prior to discharge. A chart review will be performed for all control group participants by study coordinators prior to patient discharge. Both control group participants and primary care providers (PCPs) of intervention study participants will complete questionnaires 30-60 days after hospital discharge to assess certain patient ( 10 minute questionnaire; via phone) and primary care provider ( 5 minute questionnaire via email) perceptions (Please see Aim 4 and Aim 5). A REDCap database will be used to store all questionnaire and chart review data. Readmission rates, ED visits, PCP appointment compliance, patient/ PCP perceptions will be tracked.

Three groups of research subjects will be assessed: the intervention study group, the control study group, and the PCPs of the patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include the following: enrollment in a Partners Risk Contract; agreement to participate in the study with ability to consent to enrollment, working phone number for patient contact and patient address of residence within 15 mile radius on MGH 55 Fruit Street, Boston, MA.

Exclusion Criteria:

* Exclusion criteria will include a lack of capacity to consent to enrollment ( including prisoner status) or lack of cognitive ability to complete the survey, living outside of a 15 mile radius of the MGH 55 Fruit street location and having a primary care provider outside the MGH system.

Ages: 18 Years to 109 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
30 day readmission rate | 1 month ( for 24 months)
  The number of patients readmitted within 30 days of being discharged from studied medical units during a given month/ the number of patients discharged from studied medical units during a given month

SECONDARY OUTCOMES:
Emergency Department Visit Rate | Monthly for 24 months
  The number of patient emergency department visits after discharged from studied medical units during a given month/ the number of patient emergency department visits after discharge from studied medical units during a given month
Show Rate for Primary Care Provider/ Specialist Appointments | Monthly for 24 months
  The number of primary care provider/specialist appointments attended by patients discharged from studied medical units during a given month/ The number of primary care provider/specialist appointments expected to be attended by patients discharged from studied medical units during a given month
Patient Satisfaction Post-CHW Intervention | Monthly for 24 months
  The number of patients receiving the community health worker intervention indicating they were very satisfied with CHW-patient pairing experience via questionnare/ The number of patients receiving the community health worker intervention that completed the post-CHW intervention questionnaire
Primary Care Provider Satisfaction Post CHW Intervention | Monthly for 24 months
  The number of primary care providers of patients receiving the community health worker intervention indicating they were very satisfied with CHW-patient pairing experience via questionnare/ The number of primary care providers of patients receiving the community health worker intervention that completed the post-CHW intervention questionnaire
Rates of patient depression/isolation | Monthly for 24 months
  The number of patients receiving the community health worker intervention indicating they were depressed or felt isolated via questionnare/ The number of patients receiving the community health worker intervention that completed the post-CHW intervention questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn A Carter, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kangovi S, Mitra N, Grande D, White ML, McCollum S, Sellman J, Shannon RP, Long JA. Patient-centered community health worker intervention to improve posthospital outcomes: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):535-43. doi: 10.1001/jamainternmed.2013.14327. PMID 24515422
- [Derived] Carter J, Hassan S, Walton A, Yu L, Donelan K, Thorndike AN. Effect of Community Health Workers on 30-Day Hospital Readmissions in an Accountable Care Organization Population: A Randomized Clinical Trial. JAMA Netw Open. 2021 May 3;4(5):e2110936. doi: 10.1001/jamanetworkopen.2021.10936. PMID 34014324
- [Derived] Carter J, Walton A, Donelan K, Thorndike A. Implementing community health worker-patient pairings at the time of hospital discharge: A randomized control trial. Contemp Clin Trials. 2018 Nov;74:32-37. doi: 10.1016/j.cct.2018.09.013. Epub 2018 Oct 4. PMID 30291997